CLINICAL TRIAL: NCT05849064
Title: Randomized Controlled Trial of Targeted Treatment in Older Adults Following Concussion
Brief Title: Concussion Treatment in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Anthony P. Kontos, Ph.D., Research Director, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY23020055
Record Dates: First submitted 2023-04-13; First posted 2023-05-08 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Concussion, Mild
Keywords: concussion; mild traumatic brain injury; treatment; older adults
MeSH Terms: conditions — Brain Concussion | interventions — Behavior Control

STUDY DESIGN:
Intervention Model Description: One group receives basic behavioral management strategies. The second group gets targeted treatment strategies dependent on the concussion symptoms they are expressing.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Control (Active Comparator): Participants randomized to the behavioral control group will receive standardized (i.e., all participants in this group will receive the same interventions) behavioral management strategies that include activity, hydration, nutrition, sleep, and stress management strategies.
  Interventions: Behavioral: Behavioral Control
- Targeted Intervention (Experimental): Participant receives exercises or strategies based on their clinical concussion domain given to them by their neuropsychologist: 1) Anxiety/Mood, 2)Headache/Migraine, 3)Vestibular, 4)Ocular, 5)Cognitive.
  Interventions: Behavioral: Targeted Intervention

INTERVENTIONS:
Behavioral: Behavioral Control — Participants will receive standardized behavioral management strategies for their concussion symptoms including: activity, hydration, nutrition, sleep, and stress management strategies. These strategies provide general methods to manage concussion symptoms and regulate daily activities to assist in the recovery of concussion.
  Arms: Behavioral Control
Behavioral: Targeted Intervention — Participants will be prescribed one or more interventions, tailored to their domains. Anxiety/Mood-Cog beh therapy(CBT) for maladaptive beliefs/avoidance/coping behaviors. Graded exposure/activity/relaxation exercises, cognitive restructuring. Cognitive-Accommodations for reduced work/school time/delayed deadlines, more frequent/longer cognitive rest during symptom-provoking activities. Migraine/Headache: Education, relaxation training/mindfulness based therapy. Ocular-Exercises for ocular symptoms, near point convergence, may include Brock string, pencil push-ups, fixation, saccade tracking, pursuits. Sleep-Sleep regulation/hygiene. Mindfulness-based training, morning physical activity, CBT.Vestibular-Exercises for dizziness, visual motion sensitivity, gait, imbalance that may include gaze stability, visual habituation, static and dynamic balance/gait.
  Arms: Targeted Intervention

SUMMARY:
The purpose of this study is to conduct the first randomized control trial for targeted treatments for concussion in adults 50 years or older. Participants will be enrolled at their first concussion clinical visit (V1) and their second study visit will occur after (up to 7 days) or concurrently with the participant's second concussion clinical visit, typically (but not limited to) between 21-31 days from V1.

DETAILED DESCRIPTION:
Although concussion is a common occurrence in older adults, we know little about the injury in this at-risk population. Certain management tools that might be appropriate for adolescent and young adult populations may not be appropriate for use in older adults who may have sensory, cognitive, and neuro-motor limitations. This study will help to develop initial evidence for targeted treatments for concussion in older adults. The study will utilize a two group design with permuted block random assignment to intervention and usual care/control groups. All participants will complete the following assessments at their initial and follow-up visit appointments: cognitive screening (learning, memory, language, executive functioning), concussion and mood symptom questionnaires, and neuro-motor screening. The primary outcomes for this study will be total symptom severity score (i.e., symptom burden) on the Concussion Clinical Profiles Screening (CP Screen) and Patient Global Impression of Change (PGIC). Secondary outcomes will include: Short Falls Efficacy Scale (SFES), Dizziness Handicap Inventory (DHI), Patient Health Questionnaire-9 (PHQ-9), Patient Health Questionnaire-15 (PHQ-15), Generalized Anxiety Disorder - 7 (GAD-7), Posttraumatic Stress Disorder Checklist (PCL-5), Pittsburgh Sleep Quality Index (PSQI), Neuro-Quality of Life (QOL) v2.0 - Cognition Function (Short version), Headache Impact Test (HIT-6), ID Migraine, Neck Disability Index (NDI), Vestibular Ocular Motor Screen (VOMS), Timed-Up-and-Go (TUG), Repeatable Battery for the Assessment of Neuropsychological Status (RBANS). All outcomes will be treated as continuous.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age or older
* Diagnosed concussion within the last 4 days - 12 months
* Must be recruited at their initial concussion appointment
* Ability to read/write to complete study assessments/testing

Exclusion Criteria:

* Diagnosed major psychiatric disorders other than depression/anxiety (e.g., schizophrenia)
* Diagnosed with moderate to severe brain injury or past brain surgery/malformations

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Concussion Clinical Profiles Screening (CP Screen) | Visit 1 (Baseline)
  The CP Screen is a 29 item self-report, clinical profiles based symptom inventory that measures five concussion clinical profiles: 1) anxiety/mood, 2)cognitive/fatigue, 3) migraine, 4) ocular, 5) vestibular; and two modifying factors sleep and cervical. Participants indicate on a scale of 0 (none) to 3 (severe) the level of symptom severity for each item. The CP screen yields an average factor and modifier scores, with higher scores indicative of worse symptom severity, score range is 0-87.
Concussion Clinical Profiles Screening (CP Screen) | At study completion, an average of 30 days after Visit 1
  The CP Screen is a 29 item self-report, clinical profiles based symptom inventory that measures five concussion clinical profiles: 1) anxiety/mood, 2)cognitive/fatigue, 3) migraine, 4) ocular, 5) vestibular; and two modifying factors sleep and cervical. Participants indicate on a scale of 0 (none) to 3 (severe) the level of symptom severity for each item. The CP screen yields an average factor and modifier scores, with higher scores indicative of worse symptom severity, score range is 0-87.

SECONDARY OUTCOMES:
Vestibular/Ocular Motor Screening (VOMS) | Visit 1 (Baseline)
  The VOMS assesses impairment via patient report symptom provocation following each of 5 test components (smooth pursuits, horizontal/vertical saccades, convergence, horizontal and vertical vestibular ocular reflex (VOR) and visual motor sensitivity (VMS). Patients verbally rate changes in headache, dizziness, nausea, and fogginess after each test, as well as report their baseline symptoms. Symptoms in each area are rated on scale 0 (none) to 10 (severe). Scores on any VOMS item of 2+ reflects a positive screening cut-off for vestibular and/or ocular motor impairment.
Vestibular/Ocular Motor Screening (VOMS) | At study completion, an average of 30 days after Visit 1
  The VOMS assesses impairment via patient report symptom provocation following each of 5 test components (smooth pursuits, horizontal/vertical saccades, convergence, horizontal and vertical vestibular ocular reflex (VOR) and visual motor sensitivity (VMS). Patients verbally rate changes in headache, dizziness, nausea, and fogginess after each test, as well as report their baseline symptoms. Symptoms in each area are rated on scale 0 (none) to 10 (severe). Scores on any VOMS item of 2+ reflects a positive screening cut-off for vestibular and/or ocular motor impairment.
Short Falls Efficacy Scale (SFES) | Visit 1 (Baseline)
  The SFES is a 7 item survey that measures a subject's fear and concerns about falling during normal daily life activities. Question responses are scaled from 1-4, with higher scores indicating more concern for falls. (Low concern = 7-8; Moderate concern = 9-13; High concern = 14-28).
Short Falls Efficacy Scale (SFES) | At study completion, an average of 30 days after Visit 1
  The SFES is a 7 item survey that measures a subject's fear and concerns about falling during normal daily life activities. Question responses are scaled from 1-4, with higher scores indicating more concern for falls. (Low concern = 7-8; Moderate concern = 9-13; High concern = 14-28).
Patient Health Questionnaire-9 (PHQ-9) | Visit 1 (Baseline)
  The PHQ-9 is a 9 item questionnaire that assesses the presence and severity of depression. Total score ranges from 1-27, with higher scores indicating higher level of depression. Scale is 0-4 (0=not at all, 1=several days, 2=more than half the days, 3=nearly every day).
Patient Health Questionnaire-9 (PHQ-9) | At study completion, an average of 30 days after Visit 1
  The PHQ-9 is a 9 item questionnaire that assesses the presence and severity of depression. The PHQ-9 is a 9 item questionnaire that assesses the presence and severity of depression. Total score ranges from 1-27, with higher scores indicating higher level of depression. Scale is 0-4 (0=not at all, 1=several days, 2=more than half the days, 3=nearly every day).
Patient Health Questionnaire-15 (PHQ-15) | Visit 1 (Baseline)
  The PHQ-15 comprises 15 somatic symptoms that are scored from 0 ("not bothered at all") to 2 ("bothered a lot"). Higher scores are indicative of higher levels of depression (Minimal =0-4; Low = 5-9; Medium = 10-14; High = 15=30).
Patient Health Questionnaire-15 (PHQ-15) | At study completion, an average of 30 days after Visit 1
  The PHQ-15 comprises 15 somatic symptoms that are scored from 0 ("not bothered at all") to 2 ("bothered a lot"). Higher scores are indicative of higher levels of depression (Minimal =0-4; Low = 5-9; Medium = 10-14; High = 15=30).
General Anxiety Disorder-7 (GAD-7) | Visit 1 (Baseline)
  The GAD-7 is a seven item self-reported questionnaire that measures severity of symptoms regarding anxiety. Responses are 0 = not at all, 1 = several days, 2= more than half the days, and 3 = nearly every day. Higher scores are indicative of higher anxiety (0-4 = minimal anxiety, 5-9= mild anxiety, 10-14 =moderate anxiety, 15-21 = severe anxiety.
General Anxiety Disorder-7 (GAD-7) | At study completion, an average of 30 days after Visit 1
  The GAD-7 is a seven item self-reported questionnaire that measures severity of symptoms regarding anxiety. Responses are 0 = not at all, 1 = several days, 2= more than half the days, and 3 = nearly every day. Higher scores are indicative of higher anxiety (0-4 = minimal anxiety, 5-9= mild anxiety, 10-14 =moderate anxiety, 15-21 = severe anxiety.
PCL-5 | Visit 1 (Baseline)
  The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. Responses are on a 5 point likert scale (0=not at all, 1=a little bit, 2=moderately, 3=quite a bit, 4=extremely). Overall score is total sum of 20 items with higher scores indicating higher level of PTSD (Range 0-80)
PCL-5 | At study completion, an average of 30 days after Visit 1
  The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. Responses are on a 5 point likert scale (0=not at all, 1=a little bit, 2=moderately, 3=quite a bit, 4=extremely). Overall score is total sum of 20 items with higher scores indicating higher level of PTSD (Range 0-80).
Neuro-QOL (Cognitive Function Scale - short form) | Visit 1 (Baseline)
  The cognitive function measures perceived difficulties in cognitive abilities (e.g., memory, attention, and decision making, or in the application of such abilities to everyday tasks (e.g., planning, organizing, calculating, remembering and learning). The short form contains 8 items, scored 0-5 (5=never, 4=rarely/once, 3=sometimes/2-3 times, 2=often/once a day, 1=very often/several times per day. Total scores range from 0-40. Higher scores indicate better self-reported cognitive function.
Neuro-QOL (Cognitive Function Scale - short form) | At study completion, an average of 30 days after Visit 1
  The cognitive function measures perceived difficulties in cognitive abilities (e.g., memory, attention, and decision making, or in the application of such abilities to everyday tasks (e.g., planning, organizing, calculating, remembering and learning). The short form contains 8 items, scored 0-5 (5=never, 4=rarely/once, 3=sometimes/2-3 times, 2=often/once a day, 1=very often/several times per day. Total scores range from 0-40. Higher scores indicate better self-reported cognitive function.
Dizziness Handicap Inventory (DHI) | Visit 1 (Baseline)
  The DHI is a 25 item self-reported measure that examines dizziness-related handicap. The assessment has 3 domains (functional, emotional, and physical). Participants self-report the level dizziness has impacted their abilities in the 3 domains with each domain having 9 questions (questions are answered No (0)/Sometimes(2)/Yes(4)) Item scores are summed. There is a maximum score of 100 (28 points for physical, 36 points for emotional and 36 points for functional). Minimum score is 0.
Dizziness Handicap Inventory (DHI) | At study completion, an average of 30 days after Visit 1
  The DHI is a 25 item self-reported measure that examines dizziness-related handicap. The assessment has 3 domains (functional, emotional, and physical). Participants self-report the level dizziness has impacted their abilities in the 3 domains with each domain having 9 questions (questions are answered No (0)/Sometimes(2)/Yes(4)) Item scores are summed. There is a maximum score of 100 (28 points for physical, 36 points for emotional and 36 points for functional). Minimum score is 0.
Headache Impact Test-6 (HIT-6) | Visit 1 (Baseline)
  The HIT-6 is comprised of 6 self-report items that assess frequency, severity and limitations of daily activities, fatigue, irritability, and concentration related to headaches. Items score from 6 to 13, with higher scores indicating worse severity. Scores = never = 6pts, rarely = 8 pts, sometimes = 10pts, very often = 11 pts, always = 13 points. Score range 36-78.
Headache Impact Test-6 (HIT-6) | At study completion, an average of 30 days after Visit 1
  The HIT-6 is comprised of 6 self-report items that assess frequency, severity and limitations of daily activities, fatigue, irritability, and concentration related to headaches. Items score from 6 to 13, with higher scores indicating worse severity. Scores = never = 6pts, rarely = 8 pts, sometimes = 10pts, very often = 11 pts, always = 13 points. Score range 36-78.
ID Migraine | Visit 1 (Baseline)
  The ID Migraine will be used to screen for headache symptoms. It is a 3 item screening tool designed to assess presence (yes/no) of symptoms related to headache/migraine pain. Scores range from 0-3 with clinical cut-off of 2+ indicating presence of migraines.
ID Migraine | At study completion, an average of 30 days after Visit 1
  The ID Migraine will be used to screen for headache symptoms. It is a 3 item screening tool designed to assess presence (yes/no) of symptoms related to headache/migraine pain. Scores range from 0-3 with clinical cut-off of 2+ indicating presence of migraines.
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | Visit 1 (Baseline)
  RBANS provides a brief, individually administered battery to measure cognitive decline or improvement across 5 domains (Immediate memory, visuospatial/constructional, language, attention, and delayed memory. There are total scores and indices scores, which are different depending on age and gender. Higher scores indicate better performance for all 5 domains. (<69=extremely low, 70-79=borderline, 80-89-low average, 90-109=average, 110-119=high average, 120-129=superior, 130 and higher = very superior).
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | At study completion, an average of 30 days after Visit 1
  RBANS provides a brief, individually administered battery to measure cognitive decline or improvement across 5 domains (Immediate memory, visuospatial/constructional, language, attention, and delayed memory. There are total scores and indices scores, which are different depending on age and gender. Higher scores indicate better performance for all 5 domains. (<69=extremely low, 70-79=borderline, 80-89-low average, 90-109=average, 110-119=high average, 120-129=superior, 130 and higher = very superior).
Neck Disability Index | Visit 1 (Baseline)
  Neck pain scale, each item scores 0-5 with range 0-50. Overall score out of 50 is multiplied by 100 to get a percentage. 0-20% = minimal disability, 20-40% is moderate disability, 40-60% severe disability, 60-80% = crippled, 80-100% =participants are either bed-bound or exaggerating symptoms.
Neck Disability Index | At study completion, an average of 30 days after Visit 1
  Neck pain scale, each item scores 0-5 with range 0-50. Overall score out of 50 is multiplied by 100 to get a percentage. 0-20% = minimal disability, 20-40% is moderate disability, 40-60% severe disability, 60-80% = crippled, 80-100% =participants are either bed-bound or exaggerating symptoms.
Pittsburgh Sleep Quality Index (PSQI) | Visit 1 (Baseline)
  The PSQI assesses sleep quality. It is an 19 item self-reported measure that is comprised of seven component scores: 1) subjective sleep quality, 2) sleep latency, 3) sleep duration, 4) sleep efficiency, 5) sleep disturbances, 6) sleep medication usage, and 7) daytime dysfunction. Each item is scored 0-3 (0 = very good, 1 = fairly good, 2= fairly bad, 3=very bad). Higher scores indicate more sleep dysfunction. Score range is 0-21.
Pittsburgh Sleep Quality Index (PSQI) | At study completion, an average of 30 days after Visit 1
  The PSQI assesses sleep quality. It is an 19 item self-reported measure that is comprised of seven component scores: 1) subjective sleep quality, 2) sleep latency, 3) sleep duration, 4) sleep efficiency, 5) sleep disturbances, 6) sleep medication usage, and 7) daytime dysfunction. Each item is scored 0-3 (0 = very good, 1 = fairly good, 2= fairly bad, 3=very bad). Higher scores indicate more sleep dysfunction. Score range is 0-21.
Timed-Up-and-Go | Visit 1 (Baseline)
  Walking balance test, distance of 3 meters (10 feet). Participants are timed. Participants are seated in a chair, instructed to get up, walk 3 meters (marked on floor or by cone), round the cone, return to the chair and sit back down. Participants will repeat this 3 times, and we will use the average time. < 10 second = normal, <20 seconds, good mobility, <30 second, problems/may require aid. Higher scores indicating more problems with mobility.
Timed-Up-and-Go | At study completion, an average of 30 days after Visit 1
  Walking balance test, distance of 3 meters (10 feet). Participants are timed. Participants are seated in a chair, instructed to get up, walk 3 meters (marked on floor or by cone), round the cone, return to the chair and sit back down. Participants will repeat this 3 times, and we will use the average time. < 10 second = normal, <20 seconds, good mobility, <30 second, problems/may require aid. Higher scores indicating more problems with mobility.
Patient's Global Impression of Change (PGIC) | Daily between Visit 1 and study completion, an average of 30 days
  PGIC is a self-reported assessment of change. Participants rate their impression of how much better they feel on a 7 point likert scale. It is a 1 item survey, with higher scores representing no change and associated with feeling worse. (Responses 1=much improved, 2=minimally improved, 3=no change, 4=minimally worse, 5=much worse, 6=very much worse).
Percent Back to Normal | Daily between Visit 1 and study completion, an average of 30 days
  Subject rates on a scale from 0% to 100% how much they feel like they are back to normal (before injury)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Kontos, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No